CLINICAL TRIAL: NCT06593106
Title: The CRYSTAL Study: Cryodevitalization Study for the Treatment of Early-Stage Lung Cancer
Brief Title: Cryodevitalization for the Treatment of Early Stage Lung Cancer, CRYSTAL Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Swim Across America (Other)
Responsible Party: Principal Investigator, Fabien Maldonado, Professor of Medicine, Thoracic Surgery, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC-VCTHO24099; NCI-2024-07299 (Registry Identifier: NCI, Clinical Trials Reporting Program); P30CA068485 (NIH)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Stage I Lung Cancer; Stage II Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryosurgery; Bronchoscopy; Biopsy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Patients undergo 3 freeze-thaw cycles of cryodevitalization over 30 seconds or 3, 5, or 7 minutes each during standard of care robotic bronchoscopy with biopsy on study. Patients then undergo standard of care surgical resection on study. Patients also undergo a chest x-ray on study as well as CT and tissue sample collection throughout the study.
  Interventions: Procedure: Cryosurgery; Procedure: Robotic Bronchoscopy; Procedure: Bronchoscopy with Biopsy; Procedure: Resection; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Cryosurgery — Undergo cryodevitalization
Procedure: Robotic Bronchoscopy — Undergo standard of care robotic bronchoscopy with biopsy
Procedure: Bronchoscopy with Biopsy — Undergo standard of care robotic bronchoscopy with biopsy
Procedure: Resection — Undergo standard of care surgical resection
Procedure: Chest Radiography — Undergo chest x-ray
Procedure: Computed Tomography — Undergo Computed Tomography
Procedure: Biospecimen Collection — Undergo tissue sample collection
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial studies side effects and best treatment time of cryodevitalization in treating patients with early stage (stage I or stage II) lung cancer. Cryodevitalization is a type of cryosurgery that uses a flexible probe (cryoprobe) to kill tumor cells by freezing them. It is delivered at the time of standard diagnostic robotic bronchoscopy. Using cryodevitalization may be safe, tolerable and/or effective in treating patients with early stage lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify the maximum tolerated dose (MTD) for cryodevitalization cycle duration.

OUTLINE: This is a dose-escalation study.

Patients undergo 3 freeze-thaw cycles of cryodevitalization over 30 seconds or 3, 5, or 7 minutes each during standard of care robotic bronchoscopy with biopsy on study. Patients then undergo standard of care surgical resection on study. Patients also undergo a chest radiography (x-ray) on study as well as computed tomography (CT) and tissue sample collection throughout the study.

After completion of study treatment, patients are followed up at 3 and 7 days and are then followed as clinically required per standard of care for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single pulmonary nodule with a size less than or equal to three centimeters (average long and short axis) confirmed as malignant intraprocedurally (rapid on-site evaluation with pathology assessment showing lung cancer or oligometastatic disease) without evidence of mediastinal involvement who require nodule biopsy prior to proceeding with surgical resection
* Nodules must be located in the outer 2/3 of the periphery of the lung, greater than 10 mm from the pleura and from large blood vessels or mediastinal structures to avoid injury to other visceral organs
* Patients deemed to have a surgical resection treatment option based on preoperative staging computed tomographic (CT), postoperative predicted forced expiratory volume in 1 second (FEV1) > 40% and evaluation of medical comorbidities after discussion at multidisciplinary tumor board
* Age > 18 years old

Exclusion Criteria:

* Target nodule is within the International Association for the Study of Lung Cancer (IASLC) "central zone" (including bronchial tree, major vessels, heart, esophagus, spinal cord and phrenic & laryngeal nerves), or are < 10 mm from the pleura
* Patients with an expected survival less than 6 months
* Patients with endobronchial lesions, concerning for malignancy, visualized during the initial bronchoscopic evaluation of the airways
* Patients with medically uncorrectable coagulopathy: abnormal platelet count < 100 × 10^9/L or an international normalized ratio > 1.5
* Patients with known pulmonary hypertension (PASP [pulmonary artery systolic pressure] > 50mmHg)
* Patients who are currently prescribed anticoagulants, clopidogrel, or other platelet aggregation inhibitors
* Patients with medical comorbidities deemed high-risk for surgical resection
* Pregnant women
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose for cryodevitalization cycle duration | At time of surgery
  Will implement a modified Toxicity Probability Interval design. Each dose will be modeled using a Beta-Binomial model with the prior distribution, Beta (1,1). For each dose level, a 95% credible interval for the toxicity probability will be computed.
Feasibility of bronchoscopically delivered cryodevitalization | At time of surgery
  Proportion of procedures that can be safely completed with full dose delivered
Incidence of adverse events | Up to 7 days post-cryosurgery
  Will be modeled using a Beta-Binomial model with the prior distribution, Beta (1,1). For each dose level, a 95% credible interval for the toxicity probability will be computed.

SECONDARY OUTCOMES:
Pathologic response | At time of surgical resection
  Pathologic response will be assessed comparing the confirmed devitalization zone determined by intraprocedural cone-beam computed tomography imaging (percent tumor treated by cryodevitalization) and remaining tumor viability by histopathologic examination of resected specimens.
Incidence of adverse events | From day 8 post-cryosurgery to surgical resection
  Will be modeled using a Beta-Binomial model with the prior distribution, Beta (1,1). For each dose level, a 95% credible interval for the toxicity probability will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT06593106/ICF_000.pdf